CLINICAL TRIAL: NCT05460676
Title: Reducing Distress and Tobacco Smoking in Cancer Survivors: a TDCS Telehealth Study
Brief Title: Reducing Tobacco Smoking: a Transcranial Direct Current Stimulation (TDCS) Telehealth Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00076035; 40010563 (Other: National Institute on Drug Abuse)
Record Dates: First submitted 2022-02-23; First posted 2022-07-15 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Smoking Cessation
Keywords: cigarette; smoking; cancer; anxiety; stress; tobacco; mindfulness
MeSH Terms: conditions — Smoking Cessation; Smoking; Neoplasms; Anxiety Disorders | interventions — Transcranial Direct Current Stimulation; Mindfulness

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active tDCS + Mindfulness (Experimental)
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Other: Mindfulness
- Sham tDCS + Mindfulness (Sham Comparator)
  Interventions: Other: Mindfulness; Other: Sham - Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — tDCS is noninvasive brain stimulation device that modulates brain activity by delivering a low-intensity electrical current (2.0 mA) through sponge electrodes placed on the scalp.
  Arms: Active tDCS + Mindfulness
Other: Mindfulness — Participants will follow an audio track for guided mindfulness during the stimulation.
Other: Sham - Transcranial Direct Current Stimulation (tDCS) — The tDCS device is programmed to mimic active tDCS.
  Arms: Sham tDCS + Mindfulness

SUMMARY:
The study aims to evaluate the feasibility of using Dorsolateral Prefrontal Cortex (DLPFC) Transcranial Direct Current Stimulation (tDCS) as a tool to decreasing distress and cigarette smoking. 46 participants currently smoking cigarettes, and seeking to decrease cigarette use will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* 21-75 years old
* Smoke ≥5 cigarettes per day and express interest in quitting smoking in next 30 days
* Mild to moderate distress defined as K10 scores 10-35
* Self reported previous diagnosis of cancer
* Psychotropic medication stable for ≥1 month prior to enrollment and throughout the trial, at the discretion of the study physician
* Access to a reliable internet connection, able to use mobile device, and complete online questionnaires, competent in instrumental activities of daily living
* Able to read and understand informed consent and questionnaires in English (WRAT-4 score≥85)

Exclusion Criteria:

* Inability to effectively use study-provided supplies
* Chronic non-compliance with study procedures
* Changes in health information over the course of enrollment in the study which place the participant at higher risk for an adverse event (as determined by Study Physician or Principal Investigator; e.g. medication changes, invasive procedures)
* Temporary or permanent obstructions to making contact between the electrodes and the scalp (e.g. wig that the participant is not willing to remove)
* History of traumatic brain injury, brain metastases, seizure disorder, recent (<5 years) seizure history, or a neurodegenerative disease or neurocognitive disorder associated with significant impairment (e.g. Parkinson's, Dementia)
* Current severe major depressive disorder, lifetime history of psychotic disorders or bipolar disorder type I, or current suicidal ideation
* Currently meets DSM-5 criteria for severe substance use disorder in the past 6 months for any psychoactive substance other than tobacco
* Current suicidal ideation (as determined by the MINI)
* Current use of prescription or over the counter smoking cessation medication, or primary use of non-combustible forms of nicotine/tobacco
* Currently receiving intravenous chemotherapy or radiation treatments
* Presence of metal objects in the head/neck
* Any skin disorder or skin sensitive area near stimulation locations
* Self-reported pregnancy
* Enrolled in group or individual therapy for smoking cessation that would be concurrent to intervention

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Tolerability Questionnaire (FTQ) score | 1 month
  The FTQ is a questionnaire is a 10 question survey which will be used to determine the ease and comfort of device use. Each question will be rated on a scale of 1 - 10, with 1 indicating the greatest difficulty or discomfort, and 10 indicating the greatest ease or tolerability. Questions for which the population average is greater than or equal to 5 will be deemed well tolerated.

SECONDARY OUTCOMES:
Kessler Psychological Distress Scale (K10) Score | 1 month
  K10 is a 10-item questionnaire intended to yield a global measure of distress based on questions about anxiety and depressive symptoms that a person has experienced in the most recent 4 week period. Each question is given a score between 1 (none of the time) to 5 (all of the time). The total score ranges from 10 to 50. People with scores < 20 are likely to be well, 20-24 are likely to have a mild mental disorder, 25-29 are likely to have moderate mental disorder, and > 30 are likely to have a severe mental disorder.
Weekly cigarette use | 1 month
  The timeline follow back questionnaire (TLFB) is a self report questionnaire which asks the participant to state the number of cigarettes they have smoked each day. The total number of cigarettes smoked each week will be compiled for each participant. weekly totals will be compared between the 2 arms of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Merideth A Addicott, Ph.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to chanlon@wakehealth.edu. To gain access, data requestors will need to sign a data access agreement.